CLINICAL TRIAL: NCT06030245
Title: Clostridioides Difficile Infection: Prospective Cohort Analyzing CLInic Evolution and Bacterial Clearance
Brief Title: Clostridioides Difficile Infection: Analyzing CLInic Evolution and Bacterial Clearance
Acronym: DECLIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DECLIC
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Clostridium Difficile Infections
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — additional stool samples (or Fecal Swab in the absence of stool output) to that of the initial diagnosis, as well as saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Clostridioides infection: The following procedures are specific to this test: 8 additional stool swabs (or Fecal Swab in the absence of stool output) to that of the initial diagnosis, plus four saliva swabs. Rectal swabs may cause anal irritation. The patient must also complete a stool collection form.

SUMMARY:
Clostridioides difficile (formerly Clostridium) is a bacterium found in the form of spores (resistance form) in the environment to which patients may be exposed. This bacterium used to belong to the Clostridium genus, but analysis of its 16S ribosomal RNA in 2016 led to its being distinguished from it. Once the spore has been ingested, it can germinate in vegetative form (the active form of the bacterium), taking on the appearance of a Gram-positive bacillus that will colonize the digestive microbiota. This preliminary stage of digestive colonization by the bacteria is facilitated by certain factors, notably nasogastric probing, antacids, etc. Antibiotics, for their part, disrupt the bacteria of the digestive microbiota (dysbiosis), thus facilitating the implantation of C. difficile. Certain strains (known as toxigenic) will produce the main virulence factors: toxins A (TcdA) and B (TcdB) ± a third toxin (binary toxin or CDT), and thus cause the main clinical signs of digestive infection, particularly in patients with risk factors for C. difficile infection (progressive cancer, immunodepression, etc.).

Clostridioides difficile infection (CDI) is characterized by variable clinical presentations, ranging from simple watery diarrhea without colitis, which often resolves spontaneously, to severe forms with complications such as pseudomembranous colitis, intestinal perforation or septic shock, which have a very poor prognosis.

Management of this type of CDI relies mainly on the oral administration of anti-clostridium difficile antibiotics such as fidaxomicin (FDX) or vancomycin (VAN) for 10 days, as recommended by the European ESCMID, British and American IDSA guidelines. Oral metronidazole is recommended only in the absence of availability of the first two molecules (community use). Despite this treatment, one of the main characteristics of CDI is a high recurrence rate, which can reach 25% of cases. With FDX, recurrence rates appear to be lower, especially as its administration regimen is optimized. Nevertheless, its high cost is a barrier to its wider use.

In view of the high cost to the community of treating recurrences, and the reduced quality of life of patients suffering from these recurrences, which are sometimes multiple and highly incapacitating, reducing the occurrence of recurrences is a major challenge. A better understanding of the factors leading to recurrence is therefore a prerequisite for optimizing CDI prevention and treatment strategies.

The study of colonic mucosal immunity (aimed at quantifying IgA in stools) could also contribute to a better understanding of patient progress.

All these issues surrounding CDI and its management justify the setting up of a prospective cohort for the longitudinal follow-up of infected patients, enabling us to study the digestive clearance of the bacteria according to various factors, notably the digestive microbiota and the mucosal immune response.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients hospitalized in a department of GH Paris Saint-Joseph with a microbiologically documented Clostridioides difficile infection or a microbiologically documented Clostridioides difficile recurrence.
* Patient to be treated for Clostridioides difficile infection
* French-speaking patient
* Patients who do not object to their participation in the study

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in a department of Hôpital Paris Saint-Joseph with microbiologically documented Clostridioides difficile infection or microbiologically documented recurrence of Clostridioides difficile infection, for whom treatment of Clostridioides difficile infection is to be initiated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Duration of delay between diagnosis of CDI and early or late elimination of C. difficile | Month 2
  This outcome corresponds to the kinetics of C. difficile elimination, and the time taken for the various microbiological tests (EIA, immunochromatography (ICT), culturomic and specific qPCR tests) detecting C. difficile in stools to become negative, from the day of diagnosis (i.e. before treatment was started), during the 10-day treatment period and after the end of treatment.

SECONDARY OUTCOMES:
Confronting digestive microbiota dysbiosis with C. difficile elimination kinetics | Month 2
  This outcome corresponds to the comparison in terms of number and type of digestive microbiota as a function of C. difficile elimination kinetics before treatment (at the time of diagnosis), at the end of 10 days of CDI treatment and after the end of treatment.
Impact of antibiotics prescribed for the treatment of CDI after 10 days of treatment | Day 10
  This outcome corresponds to the comparison in terms of number and type of diversity of digestive microbiota according to the type of anti-C. difficile antibiotic prescribed at the end of treatment, compared with the number and type of digestive observed at the time of diagnosis, i.e. before the start of treatment.
Determination of the form in which C. difficile persists in the digestive microbiota during treatment and after the end of treatment until it is eliminated. | Month 2
  This outcome corresponds to the type of the bacterial form (vegetative or spore-forming) that persists during and after ICD treatment by qPCR, Propidium monoazide - qPCR (PMA-qPCR) (viable or dead bacteria) and culturomics until digestive clearance of the bacteria.
Evaluation of the colonic and salivary mucosal immune response of included patients, in relation to patient progress and C. difficile elimination kinetics. | Month 2
  This outcome corresponds to the number of participants with a development of a C. difficile anti-toxin IgA response and correlation of colonic/salivary IgA levels after ICD with patient course (single, recurrent and severe forms) and C. difficile elimination kinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Assaf MIZRAHI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Fondation Hôpital Saint-Joseph, Paris, France

REFERENCES:
- [Background] Lawson PA, Citron DM, Tyrrell KL, Finegold SM. Reclassification of Clostridium difficile as Clostridioides difficile (Hall and O'Toole 1935) Prevot 1938. Anaerobe. 2016 Aug;40:95-9. doi: 10.1016/j.anaerobe.2016.06.008. Epub 2016 Jun 28. PMID 27370902
- [Background] Johnson S, Lavergne V, Skinner AM, Gonzales-Luna AJ, Garey KW, Kelly CP, Wilcox MH. Clinical Practice Guideline by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA): 2021 Focused Update Guidelines on Management of Clostridioides difficile Infection in Adults. Clin Infect Dis. 2021 Sep 7;73(5):e1029-e1044. doi: 10.1093/cid/ciab549. PMID 34164674
- [Background] van Prehn J, Reigadas E, Vogelzang EH, Bouza E, Hristea A, Guery B, Krutova M, Noren T, Allerberger F, Coia JE, Goorhuis A, van Rossen TM, Ooijevaar RE, Burns K, Scharvik Olesen BR, Tschudin-Sutter S, Wilcox MH, Vehreschild MJGT, Fitzpatrick F, Kuijper EJ; Guideline Committee of the European Study Group on Clostridioides difficile. European Society of Clinical Microbiology and Infectious Diseases: 2021 update on the treatment guidance document for Clostridioides difficile infection in adults. Clin Microbiol Infect. 2021 Dec;27 Suppl 2:S1-S21. doi: 10.1016/j.cmi.2021.09.038. Epub 2021 Oct 20. PMID 34678515
- [Background] Cornely OA, Crook DW, Esposito R, Poirier A, Somero MS, Weiss K, Sears P, Gorbach S; OPT-80-004 Clinical Study Group. Fidaxomicin versus vancomycin for infection with Clostridium difficile in Europe, Canada, and the USA: a double-blind, non-inferiority, randomised controlled trial. Lancet Infect Dis. 2012 Apr;12(4):281-9. doi: 10.1016/S1473-3099(11)70374-7. Epub 2012 Feb 8. PMID 22321770
- [Background] Guery B, Menichetti F, Anttila VJ, Adomakoh N, Aguado JM, Bisnauthsing K, Georgopali A, Goldenberg SD, Karas A, Kazeem G, Longshaw C, Palacios-Fabrega JA, Cornely OA, Vehreschild MJGT; EXTEND Clinical Study Group. Extended-pulsed fidaxomicin versus vancomycin for Clostridium difficile infection in patients 60 years and older (EXTEND): a randomised, controlled, open-label, phase 3b/4 trial. Lancet Infect Dis. 2018 Mar;18(3):296-307. doi: 10.1016/S1473-3099(17)30751-X. Epub 2017 Dec 19. PMID 29273269
- [Background] Guery B, Berger P, Gauzit R, Gourdon M, Barbut F; DAFNE study group; Dafne Study Group, Bemer P, Bessede E, Camou F, Cattoir V, Couzigou C, Descamps D, Dinh A, Laurans C, Lavigne JP, Lechiche C, Leflon-Guibout V, Le Monnier A, Levast M, Mootien JY, N'Guyen Y, Piroth L, Prazuck T, Rogeaux O, Roux AL, Vachee A, Vernet Garnier V, Wallet F. A prospective, observational study of fidaxomicin use for Clostridioides difficile infection in France. J Int Med Res. 2021 Jun;49(6):3000605211021278. doi: 10.1177/03000605211021278. PMID 34162264
- [Background] Watt M, Dinh A, Le Monnier A, Tilleul P. Cost-effectiveness analysis on the use of fidaxomicin and vancomycin to treat Clostridium difficile infection in France. J Med Econ. 2017 Jul;20(7):678-686. doi: 10.1080/13696998.2017.1302946. Epub 2017 Mar 16. PMID 28299963
- [Background] Kyne L, Warny M, Qamar A, Kelly CP. Association between antibody response to toxin A and protection against recurrent Clostridium difficile diarrhoea. Lancet. 2001 Jan 20;357(9251):189-93. doi: 10.1016/S0140-6736(00)03592-3. PMID 11213096
- [Background] Chilton CH, Crowther GS, Todhunter SL, Ashwin H, Longshaw CM, Karas A, Wilcox MH. Efficacy of alternative fidaxomicin dosing regimens for treatment of simulated Clostridium difficile infection in an in vitro human gut model. J Antimicrob Chemother. 2015 Sep;70(9):2598-607. doi: 10.1093/jac/dkv156. Epub 2015 Jun 14. PMID 26078392
- [Background] Le Monnier A, Candela T, Mizrahi A, Bille E, Bourgeois-Nicolaos N, Cattoir V, Farfour E, Grall I, Lecointe D, Limelette A, Marcade G, Poilane I, Poupy P, Kansau I, Zahar JR, Pilmis B; GMC Group. One-day prevalence of asymptomatic carriage of toxigenic and non-toxigenic Clostridioides difficile in 10 French hospitals. J Hosp Infect. 2022 Nov;129:65-74. doi: 10.1016/j.jhin.2022.05.011. Epub 2022 May 28. PMID 35640734
- [Background] Le Monnier A, Duburcq A, Zahar JR, Corvec S, Guillard T, Cattoir V, Woerther PL, Fihman V, Lalande V, Jacquier H, Mizrahi A, Farfour E, Morand P, Marcade G, Coulomb S, Torreton E, Fagnani F, Barbut F; GMC Study Group. Hospital cost of Clostridium difficile infection including the contribution of recurrences in French acute-care hospitals. J Hosp Infect. 2015 Oct;91(2):117-22. doi: 10.1016/j.jhin.2015.06.017. Epub 2015 Jul 22. PMID 26253518
- [Background] Meza-Torres J, Auria E, Dupuy B, Tremblay YDN. Wolf in Sheep's Clothing: Clostridioides difficile Biofilm as a Reservoir for Recurrent Infections. Microorganisms. 2021 Sep 10;9(9):1922. doi: 10.3390/microorganisms9091922. PMID 34576818
- [Background] Barbut F, Galperine T, Vanhems P, Le Monnier A, Durand-Gasselin B, Canis F, Jeanbat V, Duburcq A, Alami S, Bensoussan C, Fagnani F. Quality of life and utility decrement associated with Clostridium difficile infection in a French hospital setting. Health Qual Life Outcomes. 2019 Jan 11;17(1):6. doi: 10.1186/s12955-019-1081-5. PMID 30634997
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Background] Sethi AK, Al-Nassir WN, Nerandzic MM, Bobulsky GS, Donskey CJ. Persistence of skin contamination and environmental shedding of Clostridium difficile during and after treatment of C. difficile infection. Infect Control Hosp Epidemiol. 2010 Jan;31(1):21-7. doi: 10.1086/649016. PMID 19929371
- [Background] Wenisch C, Parschalk B, Hasenhundl M, Hirschl AM, Graninger W. Comparison of vancomycin, teicoplanin, metronidazole, and fusidic acid for the treatment of Clostridium difficile-associated diarrhea. Clin Infect Dis. 1996 May;22(5):813-8. doi: 10.1093/clinids/22.5.813. PMID 8722937
- [Background] Saha S, Yadav D, Pardi R, Patel R, Khanna S, Pardi D. Kinetics of polymerase chain reaction positivity in patients with Clostridioides difficile infection. Therap Adv Gastroenterol. 2021 Oct 8;14:17562848211050443. doi: 10.1177/17562848211050443. eCollection 2021. PMID 34646361
- [Background] Kyne L, Warny M, Qamar A, Kelly CP. Asymptomatic carriage of Clostridium difficile and serum levels of IgG antibody against toxin A. N Engl J Med. 2000 Feb 10;342(6):390-7. doi: 10.1056/NEJM200002103420604. PMID 10666429
- [Background] Wilcox MH, Gerding DN, Poxton IR, Kelly C, Nathan R, Birch T, Cornely OA, Rahav G, Bouza E, Lee C, Jenkin G, Jensen W, Kim YS, Yoshida J, Gabryelski L, Pedley A, Eves K, Tipping R, Guris D, Kartsonis N, Dorr MB; MODIFY I and MODIFY II Investigators. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection. N Engl J Med. 2017 Jan 26;376(4):305-317. doi: 10.1056/NEJMoa1602615. PMID 28121498
- [Background] Ahluwalia B, Magnusson MK, Ohman L. Mucosal immune system of the gastrointestinal tract: maintaining balance between the good and the bad. Scand J Gastroenterol. 2017 Nov;52(11):1185-1193. doi: 10.1080/00365521.2017.1349173. Epub 2017 Jul 12. PMID 28697651
- [Background] Nibbering B, Gerding DN, Kuijper EJ, Zwittink RD, Smits WK. Host Immune Responses to Clostridioides difficile: Toxins and Beyond. Front Microbiol. 2021 Dec 21;12:804949. doi: 10.3389/fmicb.2021.804949. eCollection 2021. PMID 34992590
- [Background] Bridgman SL, Konya T, Azad MB, Guttman DS, Sears MR, Becker AB, Turvey SE, Mandhane PJ, Subbarao P; CHILD Study Investigators; Scott JA, Field CJ, Kozyrskyj AL. High fecal IgA is associated with reduced Clostridium difficile colonization in infants. Microbes Infect. 2016 Sep;18(9):543-9. doi: 10.1016/j.micinf.2016.05.001. Epub 2016 May 24. PMID 27235197
- See also: Clostridioides difficile infection: guidance on management and treatment [Internet]. GOV.UK. 2022 — https://www.gov.uk/government/consultations/clostridioides-difficile-infection-guidance-on-management-and-treatment